CLINICAL TRIAL: NCT06061913
Title: Comparison of Breast Pump Suction Patterns in Achievement of Coming to Volume in Breast Pump-Dependent Mothers of Critically Ill Infants
Brief Title: Comparison of Breast Pump Suction Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202202805
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Insufficient Breast Milk Syndrome

STUDY DESIGN:
Intervention Model Description: This study will use a randomized control trial design with 3 arms to compare the clinical effectiveness of three different breast pump suction patterns (BPSP) on lactation outcomes among pump dependent mothers of critically ill infants who demonstrate faltering lactation on day 6-8 postpartum. Mothers identified as having faltering lactation will be randomly assigned to one of 3 groups; (1) BPSP1, (2) BPSP 2, and (3) Standard BPSP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast Pump Suction Pattern 1 (Active Comparator)
  Interventions: Behavioral: Breast Pump suction pattern
- Breast Pump Suction Pattern 2 (Active Comparator)
  Interventions: Behavioral: Breast Pump suction pattern
- Breast Pump Suction Pattern 3 (Sham Comparator)
  Interventions: Behavioral: Breast Pump suction pattern

INTERVENTIONS:
Behavioral: Breast Pump suction pattern — Mothers who have reached secretory activation and are pumping <350 mLs/day will be randomized to one of three breast pump suction patterns.

SUMMARY:
Compare effectiveness of breast pump patterns on lactation outcomes of pump dependent mothers of critically ill infants

DETAILED DESCRIPTION:
Insufficient Mothers Own Milk (MOM) has its origins during the first 14 days postpartum, a critical window that includes secretory activation (SA; milk coming in; lactogenesis II) and the achievement of coming to volume (CTV; providing 500 mLs/day of MOM by day 14 postpartum). For all lactating mothers, SA must be achieved for lactation to continue, and CTV predicts provision of MOM through to neonatal intensive care unit (NICU) discharge in preterm very low birth weight (VLBW; <1500 g birth weight) infants. For this study, we posit that alternate breast pump suction patterns (BPSP; suction rate, intensity, and rhythm) may facilitate achievement of CTV in mothers who have achieved SA, but whose daily pumped MOM volumes indicate a high risk of not achieving CTV. Therefore, the overall objective of this study is to compare the clinical effectiveness of three different breast pump suction patterns on lactation outcomes, including achievement of SA, among pump dependent mothers of critically ill infants who demonstrate faltering lactation after achievement of SA. At 6-8 days postpartum, 90 pump dependent mothers of critically ill infants who have achieved SA but demonstrate faltering lactation (<350 mLs/day pumped MOM volume), will be randomized to use one of three different BPSPs with two groups having alternative BPSPs and one group using the current practice standard for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* delivered an infant admitted to the NICU
* Intent to provide exclusive mother's own milk to their infants for the first 14 days postpartum
* Expect to be breast pump dependent for the first 14 days postpartum

Exclusion Criteria:

* Breast reduction or augmentation
* Infant not expected to survive
* Medications or maternal conditions incompatible with providing mother's own milk to a NICU infant
* Resides over 60 miles from University of Florida (UFHealth) in Gainesville, FL.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be able to bear children and produce breast milk.
Enrollment: 96 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pumped milk volume | Days 1-15 post-partum
  Daily volume of milk pumped daily

SECONDARY OUTCOMES:
Maintenance of secretory activation | Days 1-15 post-partum
  Whether sodium level < 20 is maintained
Maternal perceptions of comfort, effectiveness, efficiency, and convenience | Day 15 post-partum
  Survey will be used to collect mother's perception of comfort, efficiency, and convenience
Proportion of infant feeds consisting of mother's own milk . | Days 1 post-partum until 6 months .
  Proportion of feeds consisting of mother's own milk for first 15 days, infant discharge, as well as 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parker, PhD, Principal Investigator — University of Florida
Locations (1):
- Neonatal intensive care unit at Shands children's hospital at the Univeristy of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT06061913/Prot_000.pdf
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT06061913/ICF_001.pdf